CLINICAL TRIAL: NCT01923857
Title: A Single-Dose, Open-Label Study to Evaluate the Pharmacokinetics and Safety Profile of Androxal in Male Subjects With Impaired Renal Function
Brief Title: Evaluation of Pharmacokinetic and Safety Profile of Androxal in Male Subjects With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZA-104
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy Volunteers (Experimental): Healthy males age 18-80 with a body mass index(BMI) 25-42 mg/m^2.
  Interventions: Drug: Androxal 25 mg
- Mild Renal Impairment (Experimental): Males with mild renal impairment age 18-80 with a body mass index(BMI) 25-42 mg/m^2 (creatinine clearance 50-80 mL/min).
  Interventions: Drug: Androxal 25 mg
- Moderate Renal Impairment (Experimental): Males with moderate renal impairment age 18-80 with a body mass index(BMI) 25-42 mg/m^2 (creatinine clearance 30-50 mL/min).
  Interventions: Drug: Androxal 25 mg
- Severe renal impairment (Experimental)
  Interventions: Drug: Androxal 25 mg

INTERVENTIONS:
Drug: Androxal 25 mg
  Other Names: enclomiphene citrate

SUMMARY:
* To determine and compare the pharmacokinetics (PK) of a single dose of 25 mg Androxal in overweight male subjects with various stages of renal impairment and in volunteers with normal renal function.
* To compare the safety profile of a single dose of 25 mg Androxal in overweight male subjects with various stages of renal impairment and in volunteers with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Impaired Renal Function:

Subjects with various stages of impaired renal function must meet all of the following inclusion criteria at screening will be considered for admission to the study:

1. Speak, read, and understand English or Spanish and is willing and able to provide written informed consent on an Institutional Review Board (IRB)-approved form prior to the initiation of any study procedures;
2. Male, between the ages of 18 and 80 years with Body Mass Index (BMI) between 25 and 42, inclusive, are preferred.
3. Subjects must meet the criteria of mildly (creatinine clearance 50-80 mL/min) or moderately (creatinine clearance 30-50 mL/min) impaired renal function. The Investigator will assess the renal impairment category of each subject. Substantiation for the diagnosis must be indicated in source documents; (See Appendix B)
4. Subjects must have evidence of stable renal impairment as determined by the Investigator (See Section 9.3.2, Day -1)
5. If on medications for treatment of the complications of renal disease, and other concomitant chronic illnesses, subjects must have been taking the medications at a stable dose for at least 10 days prior to the first Androxal dosing date and are then to be continued at the same dose for the duration of the study. The medications must be recorded in source documents;
6. Subject is willing to remain in the clinic for the screening visit (approximately 1 day for the screening visit) and for the treatment visit (approximately 3 days);
7. Non-smokers are preferred, but as this is a very restricted population light to moderate smoking will be allowed (no more than 10 cigarettes/day);
8. Must be able to swallow gelatin capsules;

Subjects with Normal Renal Function:

Healthy volunteers meeting all of the following inclusion criteria at screening will be considered for admission to the study:

1. Speak, read, and understand English or Spanish and is willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures;
2. Male, between the ages of 18 and 60 years with Body Mass Index (BMI) between 25 and 39, inclusive;
3. Creatinine clearance > 80 mL/min;
4. Subjects in the control group, generally matched for age and BMI to patients enrolled in the test groups: should be ± 20 years of the mean of mildly and moderately renally impaired subjects included in the study and ± 20% of the average BMI of mildly and moderately renally impaired subjects;
5. No significant abnormal findings at the screening physical examination as evaluated by the Investigator;
6. Normal laboratory values or clinically insignificant findings at screening as determined by the Investigator;
7. Subject is willing to remain in the clinic for the screening visit (approximately 1 day for the first screening visit) and for the treatment visit (approximately 3 days);
8. No tobacco (nicotine products) use for at least three (3) months prior to the study;
9. Must be able to swallow gelatin capsules

Exclusion Criteria:

Subjects with Impaired Renal Function

Subjects with various stages of impaired renal function meeting any of the following exclusion criteria at screening will not be enrolled in the study:

1. Known hypersensitivity to Clomid;
2. Subjects with clinically significant abnormal liver function as determined by the Investigator;
3. Subjects who are treated with dialysis;
4. A physical illness within three (3) months of the study that would interfere with the study as determined by the Investigator;
5. Participation in a clinical trial with investigational medication within four (4) weeks prior to study medication administration;
6. A hematocrit >54% or a hemoglobin >17 g/dL. (Sponsor may approve enrollment of subjects with hemoglobin up to 17.5 g/dL if the subject is at a location with high elevation).
7. An acute illness within five (5) days of study medication administration;
8. Uncontrolled hypertension based on the Investigator's assessment at baseline. Subjects treated for Type II diabetes will be allowed into the study. Newly diagnosed diabetics need to be treated for at least 48 hours before being enrolled into the study.
9. Positive urine drug or infectious disease screen at the screening visit based on laboratory testing;
10. A mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude, as determined by the Investigator;
11. History of venous thromboembolic disease (e.g. deep vein thrombosis or pulmonary embolism);
12. History of myocardial infarction, unstable angina, symptomatic heart failure, ventricular dysrhythmia, or known history of corrected QT interval (QTc) interval prolongation;
13. The use of prohibited concomitant medications:

    * Drugs that may interfere with cytochrome P450 2D6 (CYP2D6) activity must cease for 7 days prior to first dose of study drug;
14. An employee or family member of an employee of the study site or the Sponsor.

Subjects with Normal Renal Function:

Healthy volunteers meeting any of the following exclusion criteria at screening will not be enrolled in the study:

1. Known hypersensitivity to Clomid;
2. Abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant by the Investigator;
3. Subjects with clinically significant abnormal liver function as determined by the Investigator;
4. Subject with a significant organ abnormality or disease as determined by the Investigator;
5. A physical illness within three (3) months of the study that would interfere with the study as determined by the Investigator;
6. Uncontrolled hypertension based on the Investigator's assessment at baseline. Subjects treated for Type II diabetes will be allowed into the study. Newly diagnosed diabetics need to be treated for at least 48 hours before being enrolled into the study.
7. A hematocrit >54% or a hemoglobin >17 g/dL. (Sponsor may approve enrollment of subjects with hemoglobin up to 17.5 g/dL if the subject is at a location with high elevation).
8. Participation in a clinical trial with investigational medication within four (4) weeks prior to study medication administration;
9. An acute illness within five (5) days of study medication administration;
10. A mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude, as determined by the Investigator;
11. History of venous thromboembolic disease (e.g. deep vein thrombosis or pulmonary embolism);
12. History of myocardial infarction, unstable angina, symptomatic heart failure, ventricular dysrhythmia, or known history of QTc interval prolongation;
13. The use of prohibited concomitant medications:

    * Drugs that may interfere with CYP2D6 activity must cease for 7 days prior to first dose of study drug;
14. An employee or family member of an employee of the study site or the Sponsor.
15. Positive urine drug or infectious disease screen at the screening visit based on laboratory testing;

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | 24 hours
  Pharmacokinetic parameters calculated as a ratio in subjects with mild or moderate renal impairment to normal after a single dose of 25 mg Androxal.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Miami, Florida
  - Minneapolis, Minnesota

REFERENCES:
- See also: Sponsor Web Site — http://www.reprosrx.com